CLINICAL TRIAL: NCT01763281
Title: Imaging the Effect of Experimental Stress on Small and Large Bowel Water During Fructose Absorption
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: E12072012SCS
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRH (Active Comparator): 100 microgram bolus of Cortisol Releasing Hormone intravenous injection given at a 20 minutes prior to Fructose drink during one of the two visits.
  The placebo comparator will be 0.9% saline (1ml) bolus injection given intravenously at the same time point during one of the two visits
  Interventions: Drug: CRH
- Normal Saline (0.9%) (Placebo Comparator): 100 microgram bolus of Cortisol Releasing Hormone intravenous injection given at a 20 minutes prior to Fructose drink during one of the two visits.
  The placebo comparator will be 0.9% saline (1ml) bolus injection given intravenously at the same time point during one of the two visits
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CRH
  Other Names: Generic name: Corticorelin trifluroacetate; Proprietary name: CRH Ferring
  Arms: CRH
Drug: Placebo
  Other Names: Normal Saline (0.9%)
  Arms: Normal Saline (0.9%)

SUMMARY:
The investigators have been developing new, non-invasive magnetic resonance imaging (MRI) techniques to image the small bowel. Building on those studies the investigators want to study, in healthy volunteers, the effects of stress on the water content of the small bowel following ingestion of fructose. This is important because in Irritable Bowel Syndrome (IBS), there seems to be a strong association of stress and anxiety with the severity of the disease. Many IBS patients complain of food intolerances and recent studies have suggested that food with high content of fructose can worsen symptoms of IBS. The investigators will carry out a study in which the investigators will induce a moderate state of stress in healthy volunteers using an injection of corticotrophin release hormone, feed them a drink containing fructose and image their bowel at intervals using MRI. Improving our understanding of the effects of stress and fructose on small bowel physiology will help us to understand better some aspects of the symptoms such as bloating, altered bowel habit and abdominal discomfort, experienced by the IBS patients and to guide therapy. The investigators hypothesize that the effect of CRH will cause significant decrease in small bowel water content (SBWC) and a faster small bowel transit with increased malabsorption following consumption of fructose.

DETAILED DESCRIPTION:
A single centre, randomized cross over study consisting a screening visit and 2 test days which will be approximately 7 days apart. The participants will receive 1g unlabelled lactose ureide in a glass of water 3 times a day on the day before the study day to induce the enzyme activity in the colonic bacteria. The participants (20 healthy volunteers) will have a baseline scan in a 1.5T MRI scanner before having a small intravenous needle inserted into their forearm. Following this procedure, the participant will have another scan before being given either a saline (0.9% NaCl) or 100microgram of CRH intravenous injection. 40g of fructose and 500mg of labeled C-13 lactose ureide dissolved in water with pure lime juice as flavorant made up to 500mL will be given to the participants. They will then have a serial scanning of the abdomen at 30-60 minutes interval for 5 hours post prandially. Salivary cortisol will be collected after every MRI scans. Participants will also be asked to blow into the hydrogen breath machine and to fill in symptom questionnaire following each MRI scans. Further breath collections for orocaecal transit time will be collected initially every 10 minutes for the first hour and 15 mins until the end of the study day. Mouthwash will be used before initial breath test collection. This procedure will be repeated again on the 2nd test day with either a saline or 100microgram of CRH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers who are 18-60 years old
* Age ≥ 18 and ≤ 60 year at pre-study investigation.
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2
* Able to give voluntary informed consent to participate in the study
* Able to understand the requirements of the study including anonymous publication and free to cooperate with the study procedures

Exclusion Criteria:

* Lactose intolerance
* Any history of serious acute or chronic illness especially gastrointestinal
* Any history of Raynaud's syndrome or impairment of circulation
* Any history of heart or lung disease
* Pregnancy or breastfeeding
* Smoking
* Unsuitable for MRI scanning (i.e. have metal implants or pacemaker)
* Regular medication interfering with gastrointestinal function, opiates or constipating drugs
* Substance abuse
* Have taken part in any other clinical study within the previous 3 months
* Previous gastrointestinal surgery
* Use of medication which interferes with study measurements or bowel motility (as judged by the study physician) such as antibiotics in the 2 weeks before pre-study examination or probiotics.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Effect of CRF on area under curve volume versus time curve for small bowel water | 430 minutes in total
  Magnetic Resonance Imaging will be used to measure small bowel water at 30-60 minutes intervals for a total of 430 minutes
Effect of CRF on increase in volume of gas in colon at 255 minutes | 15 minutes
  Magnetic resonance imaging will be used to assess colonic gas at 255 minute time point

SECONDARY OUTCOMES:
Gastric Emptying | 430 minutes
  Magnetic Resonance Imaging will be used to assess gastric emptying at 30-60 minute intervals for a total of 430 minutes
small bowel transit time using lactose C-13 ureide | 430 minutes
  Unlabelled lactose ureide 1g x3/day will be given 24 hours prior to study day. They will then be given 500mg 13C labelled lactose ureide on the study day and breath collections every 10 minutes initially for 1 hour and every 15 minute for subsequent hours
Ascending colon volume | 430 minutes
  Ascending colon volumes will be assessed using the Magnetic Resonance Imaging technique at 30-60 minute intervals
Volume of gas in colon | 430 minutes
  Volume of gas in colon will be assessed using the Magnetic Resonance Imaging technique at 30-60 minute intervals
salivary cortisol level versus small bowel water content | 430 minutes
  Saliva samples will be collected at the 30-60 minute intervals (as per the magnetic resonance imaging scans for small bowel water content)
Correlating symptom scores on the study day and Bristol Stool diary | 7 days
  Stool diary to be collected for a week

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, MD FRCP, Study Chair — University of Nottingham; Ching Lam, MBchB MRCP, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Sir Peter Mansfield Magnetic Resonance Centre, University of Nottingham, Nottingham
  - NIHR Nottingham Digestive Diseases Biomedical Research Unit, Nottingham

REFERENCES:
- [Derived] Murray KA, Lam C, Rehman S, Marciani L, Costigan C, Hoad CL, Lingaya MR, Banwait R, Bawden SJ, Gowland PA, Spiller RC. Corticotropin-releasing factor increases ascending colon volume after a fructose test meal in healthy humans: a randomized controlled trial. Am J Clin Nutr. 2016 May;103(5):1318-26. doi: 10.3945/ajcn.115.125047. Epub 2016 Apr 20. PMID 27099247